CLINICAL TRIAL: NCT03397225
Title: A Lifestyle Intervention for Type 2 Diabetes Patients in Kuwait and Its Impact on Glycaemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Mai Alhazzaa, MD, PhD student, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13/53
Record Dates: First submitted 2017-12-29; First posted 2018-01-11 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Noninsulin-Dependent; Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): The lifestyle intervention, including educational sessions were given to the intervention group of diabetes patients. The educational sessions were scheduled every two weeks and a total of four sessions was provided to the intervention group, the session held in the lecture room at the polyclinic. Also, they were received two individual sessions including dietary and physical activity advice during the consultation session in the diabetic clinic at the beginning and at the end of the study.
  Interventions: Behavioral: Lifestyle intervention
- Control group (Active Comparator): Lifestyle intervention, including individual lifestyle consultation, including dietary and physical activity consultation at the beginning and the end of the study, two sessions. This is done after the screening of the participants in the diabetic clinic at the beginning and at the end of the study.
  Interventions: Behavioral: Lifestyle intervention
- Anonymous data (No Intervention): The patients, n = 60, were recruited randomly and anonymously from the same diabetes clinic, and the HbA1c data was taken from the anonymous patients at two points over the 12-month study duration.

INTERVENTIONS:
Behavioral: Lifestyle intervention — The educational sessions and individual sessions including dietary management and physical activity advices.
  Other Names: Dietary and physical activity advices
  Arms: Control group; Intervention group

SUMMARY:
This was an unblinded, randomised controlled study, the purpose of which was to investigate the impact of a structured health education intervention on the glycaemic control of Type 2 diabetes patients within a Kuwaiti cultural context.

DETAILED DESCRIPTION:
The control group continued to receive routine clinical advice, in addition to the individual session. The intervention group was enrolled in a structured group-based educational program for the duration of the study (12 months). Physical, physiological and biochemical outcome measures were assessed at baseline and then at a 12-month follow up. The total duration of the study, including the recruitment, the screening, the pilot study, the educational sessions and the follow-up, was 14 months altogether, from December 2014 to February 2016. The study consisted of the following three phases.

* Phase 1: included the initial recruiting of diabetes patients at an Al-Rehab polyclinic and the baseline assessment of their medical, dietary and physical activity history, in addition to the biochemical assessment.
* Phase 2 (pilot study): Five patients were chosen from the recruited patients for a pilot study to be monitored for one whole month (30 days) in order to evaluate the lifestyle intervention's safety, its compliance to the educational sessions, and anticipated barriers and results. Recruitment continued during the pilot study.
* Phase 3 (main study): This phase was based on recommending lifestyle intervention to the intervention group of diabetes patients. The educational sessions were scheduled every two weeks and a total of four sessions was provided. Both intervention and control groups were received individual sessions at the beginning and at the end of the study.

Later, there was a follow up of the intervention and the control groups at the end of the study, to measure the intervention's effectiveness and evaluate the results.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, treated with diabetes medications but not on insulin only, and who had other chronic diseases associated with diabetes, such as hypertension and hyperlipidaemia

Exclusion Criteria:

* History of major disabilities such as cardiovascular disease (CVD), an inability to walk, cancer, and Chronic Obstructive Pulmonary Diseases (COPD).

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2015-01-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 months
  Diabetes control

CONTACTS AND LOCATIONS:
Overall Officials: Mai Alhazzaa, Md, PhD, Principal Investigator — University of Reading
Locations (2):
- Al-Rehab polyclinic, Kuwait City, Farwaniyah, Kuwait
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- See also: The reference is related to the background of the study — https://www.ncbi.nlm.nih.gov/pubmed/20876408